CLINICAL TRIAL: NCT01699386
Title: Growth of Infants Fed an Elemental Medical Food
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH73
Record Dates: First submitted 2012-10-02; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Infants
MeSH Terms: interventions — pregestimil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Study Formula (Active Comparator): protein hydrolysate formula
  Interventions: Other: Control Study Formula
- Experimental Study Formula (Experimental): free-amino acid-based medical food
  Interventions: Other: Experimental Study Formula

INTERVENTIONS:
Other: Control Study Formula — feed as lib
  Other Names: protein hydrolysate formula; Nutramigen
  Arms: Control Study Formula
Other: Experimental Study Formula — feed as lib
  Other Names: free-amino acid-based medical food; EleCare
  Arms: Experimental Study Formula

SUMMARY:
Effects on weight will be monitored in healthy infant subjects consuming assigned infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, healthy infant
* Gestational age of 37 to 42 weeks
* Birth weight of 2500 grams or greater
* Age between birth and 9 days of age
* Parents agree to not administer mineral or vitamin supplements during the study period
* Parents agree to feed study formula exclusively for the duration of the study

Exclusion Criteria:

* Maternal, fetal or perinatal history which may have adverse effects on growth
* Multiple birth

Max Age: 9 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 1999-04; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Weight | 14 days of age to 112 days of age
  weight gain during the study period

SECONDARY OUTCOMES:
Anthropometric Measurements | 14 days of age to 112 days of age
  length, head circumference, and length gain
GI Tolerance | At visits 14 and 28
  daily stool number, stool consistency, formula intake
Lab Measurement | At 112 day visit
  serum albumin

CONTACTS AND LOCATIONS:
Overall Officials: Marlene W Borschel, PhD, RD, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - T&W Research, Little Rock, Arkansas
  - University of Iowa, Iowa City, Iowa

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765